CLINICAL TRIAL: NCT02620358
Title: Two Opposite Strategies of Weaning From Mechanical Ventilation: High Work of Breathing Versus Low Work of Breathing
Brief Title: Two Opposite Strategies of Weaning From Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Althaia Xarxa Assistencial Universitària de Manresa (Other)
Collaborators: Hospital Universitario Reina Sofia de Cordoba (Other Government); Hospital of Navarra (Other); Hospital Universitario Marqués de Valdecilla (Other); Hospital de Toledo (Unknown); Hospital del Mar (Other); Hospital de Mataró (Other); Hospital de Sabadell (Other); Hospital de Sant Joan Despí Moisès Broggi (Other); Consorci Sanitari de Terrassa (Other); Hospital Mutua de Terrassa (Other); Hospital Universitari Joan XXIII de Tarragona. (Other); Hospital General Universitario de Alicante (Other); Hospital General Universitario Elche (Other); Hospital Clínico Universitario de Valencia (Other); Complejo Hospitalario Universitario de Badajoz (Other); Complejo Hospitalario Universitario de Santiago (Other); Complexo Hospitalario de Ourense (Other); Complejo Hospitalario Universitario de Vigo (Other); Hospital de Henares (Other); Hospital General Universitario Gregorio Marañon (Other); Hospital Universitario Rey Juan Carlos (Other); Hospital Universitario Infanta Cristina (Other); Hospital Universitario Central de Asturias (Other); Hospital General Universitario Morales Meseguer (Other); Hospital Universitario Araba (Other); Hospital Universitario de Canarias (Other); Complejo Hospitalario de Caceres (Other); Hospital de Sagunto (Other); Hospital de Granollers (Other); Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Carles Subirà Cuyàs, Physician, Althaia Xarxa Assistencial Universitària de Manresa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEIC 15/82
Record Dates: First submitted 2015-11-20; First posted 2015-12-03 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Weaning Failure
Keywords: Mechanical Ventilation; Weaning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Work of Breathing (Experimental): If patient has weaning criteria, a Spontaneous Breathing Trial (SBT) with T Tube for 2 hours will be done.
  The patient will be extubated after the SBT if he has no criteria of SBT failure.
  Interventions: Other: T Tube for 120 minuts
- Low Work of Breathing (Experimental): If patient has weaning criteria a Spontaneous Breathing Trial (SBT) with Pressure Support Ventilation of 8 cmH2O for 30 minutes will be done.
  The patient will be extubated after the SBT if he has no criteria of SBT failure.
  Interventions: Other: Pressure Support Ventilation of 8 cmH2O for 30 minutes

INTERVENTIONS:
Other: T Tube for 120 minuts — Spontaneous Breathing Trial using T Tube for 120 minutes.
  Arms: High Work of Breathing
Other: Pressure Support Ventilation of 8 cmH2O for 30 minutes — Spontaneous Breathing Trial using Pressure Support Ventilation of 8 cmH2O for 30 minutes
  Arms: Low Work of Breathing

SUMMARY:
This study compares two opposite strategies of weaning from Mechanical Ventilation. One of them is Low Pressure Support Ventilation during 30 minutes and the other is T-Tube for 2 hours. The aim of the study is to know witch one has a higher successful extubation rate.

DETAILED DESCRIPTION:
The final stage of weaning from Mechanical Ventilation is known as Spontaneous Breathing Test (SBT). Some studies in the last 20 years have compared different strategies of weaning.

The SBT using T-Tube versus Low Pressure Support Ventilation (PSV) for 2 hours didn't show differences in successful extubation.

No difference in successful extubation rate were seen with the T-Tube for 30 or 120 minutes, or the Low PSV for 30 minutes or 2 hours For this reason the actual guidelines recommend to use T-Tube or Low PSV from 30 minutes to 2 hours with the same level of evidence.

Nevertheless, no studies have compared two opposite strategies like T-Tube for 2 hours (High work of breathing) versus Low PSV for only 30 minutes (Low work of breathing). Whereas the high work of breathing approach can be more specific for detecting more fitted patients, the low work of breathing method may reduce fatigue during SBT allowing more patients to be extubated.

We have designed a prospective, multicentric controlled and randomized study to compare this two opposite strategies of weaning: T-Tube for 120 minutes versus PSV 8 cmH2O for 30 minutes.

When patients show weaning criteria the randomly assigned SBT will be done.

We consider weaning criteria:

* Adequate cough
* Not too many respiratory secretions.
* Primary pathology solved.
* Clinical stability: Heart Rate (HR) < 140 bpm, Systolic Blood Pressure (SBP) 90-160 mmHg.
* Correct oxygenation: SatO2 > 90% with FiO2 < 0,4.
* Correct ventilatory pattern: Respiratory rate (RR) < 35 pm, Maximal Inspiratory Pressure (MIP) < -20 cmH2O, Tidal volume (TV) > 10 ml/kg, RR/TV < 100 pm/l.
* Adequate level of consciousness

Patients who succeed SBT will be extubated. Patients who fail SBT will be reconnected to the ventilator in the previous modality. These patients won't be randomized in future SBT.

We consider SBT failure:

Subjective Index:

* Neurological: Agitation or anxiety, Low level of consciousness.
* Increased work of breathing: accessory muscle use, dyspnea.

Objective Index:

* Hypoxemia: PaO2 < 60 mmHg or SatO2 < 90% with FiO2 > 50%.
* Tachypnea: RR > 35 pm.
* Hemodynamic instability: HR > 140 bpm, SBP > 180 mmHg, Arrhythmia.

Extubation failure will be registered within the first 72 hours after extubation.

We consider extubation failure:

* Respiratory acidosis: pH < 7,32, PaCO2 > 45 mmHg.
* Hypoxemia: SatO2 < 90% or PaO2 < 60 mmHg with FiO2 > 0,5.
* Deteriorating level of consciousness, Glasgow Coma Scale < 13.
* Uncontrolled agitation.
* Signs of fatigue.

Treatment of extubation failure will be decided by the attending physician: Reintubation, High Flow Oxygen therapy or Non Invasive Ventilation.

Reintubated patients won't be randomized in future SBT.

An interim analysis will be done when half of the simple is recruited.

Successful extubation will be analyzed by Kaplan-Meier survivial curves and logistic multivariable analysis with confounding variables.

ELIGIBILITY:
Inclusion Criteria:

* More tan 18 years old
* More tan 24 hour of Mechanical Ventilation ready for weaning

Exclusion Criteria:

* Tracheostomy
* Non reintubation orders

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1190 (Actual)
Dates: Start 2016-01-11 (Actual); Primary Completion 2017-03-28 (Actual); Study Completion 2017-03-28 (Actual)

PRIMARY OUTCOMES:
Succesful extubation rate | 72 hours
  Rate of succesful extubation after one of the weaning strategy

SECONDARY OUTCOMES:
ICU Length of Stay | 3 month
  Define the ICU Length os Stay of each group
Hospital Length of Stay | 3 month
  Define the Hospital Length of Stay of each group
Mortality | 3 month
  Definte mortality rate of each group
Reintubation rate | 72 hours
  Rate of reintubation in each group the first 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Fernandez Rafael, MD, Study Director — Althaia Xarxa Assistencial Manresa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Perren A, Domenighetti G, Mauri S, Genini F, Vizzardi N. Protocol-directed weaning from mechanical ventilation: clinical outcome in patients randomized for a 30-min or 120-min trial with pressure support ventilation. Intensive Care Med. 2002 Aug;28(8):1058-63. doi: 10.1007/s00134-002-1353-z. Epub 2002 Jul 13. PMID 12185425
- [Background] Esteban A, Anzueto A, Alia I, Gordo F, Apezteguia C, Palizas F, Cide D, Goldwaser R, Soto L, Bugedo G, Rodrigo C, Pimentel J, Raimondi G, Tobin MJ. How is mechanical ventilation employed in the intensive care unit? An international utilization review. Am J Respir Crit Care Med. 2000 May;161(5):1450-8. doi: 10.1164/ajrccm.161.5.9902018. PMID 10806138
- [Result] Brochard L, Rauss A, Benito S, Conti G, Mancebo J, Rekik N, Gasparetto A, Lemaire F. Comparison of three methods of gradual withdrawal from ventilatory support during weaning from mechanical ventilation. Am J Respir Crit Care Med. 1994 Oct;150(4):896-903. doi: 10.1164/ajrccm.150.4.7921460.
- [Result] Esteban A, Alia I, Tobin MJ, Gil A, Gordo F, Vallverdu I, Blanch L, Bonet A, Vazquez A, de Pablo R, Torres A, de La Cal MA, Macias S. Effect of spontaneous breathing trial duration on outcome of attempts to discontinue mechanical ventilation. Spanish Lung Failure Collaborative Group. Am J Respir Crit Care Med. 1999 Feb;159(2):512-8. doi: 10.1164/ajrccm.159.2.9803106. PMID 9927366
- [Result] Esteban A, Alia I, Gordo F, Fernandez R, Solsona JF, Vallverdu I, Macias S, Allegue JM, Blanco J, Carriedo D, Leon M, de la Cal MA, Taboada F, Gonzalez de Velasco J, Palazon E, Carrizosa F, Tomas R, Suarez J, Goldwasser RS. Extubation outcome after spontaneous breathing trials with T-tube or pressure support ventilation. The Spanish Lung Failure Collaborative Group. Am J Respir Crit Care Med. 1997 Aug;156(2 Pt 1):459-65. doi: 10.1164/ajrccm.156.2.9610109. PMID 9279224
- [Result] Esteban A, Anzueto A, Frutos F, Alia I, Brochard L, Stewart TE, Benito S, Epstein SK, Apezteguia C, Nightingale P, Arroliga AC, Tobin MJ; Mechanical Ventilation International Study Group. Characteristics and outcomes in adult patients receiving mechanical ventilation: a 28-day international study. JAMA. 2002 Jan 16;287(3):345-55. doi: 10.1001/jama.287.3.345. PMID 11790214
- [Derived] Subira C, Hernandez G, Vazquez A, Rodriguez-Garcia R, Gonzalez-Castro A, Garcia C, Rubio O, Ventura L, Lopez A, de la Torre MC, Keough E, Arauzo V, Hermosa C, Sanchez C, Tizon A, Tenza E, Laborda C, Cabanes S, Lacueva V, Del Mar Fernandez M, Arnau A, Fernandez R. Effect of Pressure Support vs T-Piece Ventilation Strategies During Spontaneous Breathing Trials on Successful Extubation Among Patients Receiving Mechanical Ventilation: A Randomized Clinical Trial. JAMA. 2019 Jun 11;321(22):2175-2182. doi: 10.1001/jama.2019.7234. PMID 31184740